CLINICAL TRIAL: NCT00504062
Title: A Randomized, Open-label, Parallel-group, 6 Week Treatment, Multi-center, Phase III Study to Investigate the Efficacy and Safety of 100ug and 200ug Twice Daily of Budesonide Turbuhaler® and 50ug and 100umg Twice Daily of Fluticasone Diskus® in Japanese Children With Bronchial Asthma Aged 5-15
Brief Title: Open-label, Safety and Efficacy Study of Pulmicort® Turbuhaler® in Japanese Children With Bronchial Asthma
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: D5254C00769
Record Dates: First submitted 2007-07-17; First posted 2007-07-19 (Estimated); Last update posted 2011-08-24 (Estimated); Status verified 2011-08

CONDITIONS: Asthma
Keywords: asthma; bronchial
MeSH Terms: conditions — Asthma | interventions — Budesonide; Fluticasone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: budesonide
  Other Names: Pulmicort® Turbuhaler®
Drug: fluticasone

SUMMARY:
To investigate the effect and safety of budesonide Turbuhaler® 100 μg/dose and 200 μg/dose twice daily for 6 weeks in Japanese children with bronchial asthma aged 5 years to 15 years old in need for inhaled glucocorticosteroid treatment. To compare the efficacy of budesonide Turbuhaler® 100 μg/dose and 200 μg/dose twice daily for 6 weeks to that of fluticasone Diskus® 50 μg/dose and 100 μg/dose twice daily for 6 week.

ELIGIBILITY:
Inclusion Criteria:

* Provision of signed written informed consent by patient's legal representative; when possible a signed written informed consent should be obtained from the patient themselves
* Patients diagnosed as having bronchial asthma regardless of type of asthma i.e. perennial or seasonal, atopic or non-atopic
* Males/females 5-15 yrs old who are able to experience to inhale with turbuhaler and diskus. the investigator will check whether the patient can inhale appropriately using training devises and "Turbuhaler trainer"
* Patients with bronchial asthma who require treatment with inhaled steroids (patients with drug therapy, in whom asthma is poorly controlled)
* Patients who are already treated with inhaled GCS should have at least 3 months prehistory of asthma before obtaining the written informed consent

Exclusion Criteria:

* Use of regular(more than 3 days) systemic (oral, intravenous or intramuscular) steroids within 30 days before the observation period
* The daily dose of inhaled GCS within 30 days before the observation period for the patients who are already treated with inhaled GCS is beyond fluticasone propionate (FP) 200 µg/day or beclomethasone dipropionate (BDP) 200 μg/day.
* Respiratory infections that, in the opinion of the investigator(s), may affect the efficacy evaluation e.g. lower airways infection such as pneumonia, infection with no available effective antimicrobial drugs or with deep seated mycosis within 30 days before the observation period.
* Concurrent serious diseases of liver, kidney, heart or other complications which, in the opinion of the investigator(s), may either put the patient at risk because of participation in the study, or may influence the results of the study, or the patient's ability to participate in the study
* Contra-indications (e.g., known or suspected allergy) to budesonide, fluticasone or lactose contained in the investigational product
* Participation in another clinical study within 12 weeks prior to the observation period or during the study
* Previous enrolment in the present study
* Current use of budesonide turbuhaler
* Pregnancy or possible pregnancy, or planning to be pregnant during the study period
* Patients whose legal representative/caregiver is involved in the planning and conduct of the study (applies to both AstraZeneca staff or staff at the study site)
* Other subjects who are considered inappropriate to participate in this study as judged by the investigator

Ages: 5 Years to 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 240 (Actual)
Dates: Start 2006-10; Study Completion 2007-10 (Actual)

PRIMARY OUTCOMES:
To investigate the effect of budesonide Turbuhaler® 100 μg/dose twice daily and 200 μg/dose twice daily for 6 weeks in Japanese children with bronchial asthma aged 5 years to 15 years old in need for inhaled glucocorticosteroid treatment | 6 weeks

SECONDARY OUTCOMES:
To investigate the safety of budesonide Turbuhaler 100 μg/dose twice daily and 200 μg/dose twice daily for 6 weeks in Japanese children with bronchial asthma aged 5 years to 15 years old in need for inhaled glucocorticosteroid treatment | 6 weeks
To compare the efficacy of budesonide Turbuhaler 100 μg/dose twice daily and 200 μg/dose twice daily for 6 weeks to that of fluticasone Diskus® 50 μg/dose twice daily and 100 μg/dose twice daily for 6 weeks | 6 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Lars-Goran Carlsson, MD, Study Director — AstraZeneca R&D Lund
Locations (1):
- Research Site, Takizawa, Iwate, Japan